CLINICAL TRIAL: NCT00155311
Title: The Regulation of Osteoprotegerin by Mechanical Stimulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 9361700741
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Malocclusion
Keywords: orthodontic tooth movement; OPG; RANKL
MeSH Terms: conditions — Malocclusion | interventions — Orthodontics

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- days after treatment (Experimental): different days after orthodontic treament, samples will be taken.
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: orthodontic treatment

SUMMARY:
To test whether levels of OPG can be changed during orthodontic treatment. Alveolar bone samples will be collected from partially impacted third molars after orthodontic uprighting for different period of time in volunteers. In situ hybridization and immunohistochemistry analysis for OPG and RANKL will reveal their roles in this physiological process.

DETAILED DESCRIPTION:
Long treatment time is a major factor causing high fee for orthodontic treatment. Patients would have dental caries or periodontitis resulted from improper oral hygiene care during this long treatment period. Therefore, how to speed up the tooth movement which determines the duration of orthodontic treatment, can help more people to obtain good occlusion and esthetics. Orthodontic force on tooth induces bone resorption on the compression side and bone deposition on the tension side, thus bone remodels and then tooth moves. Bone resorption is a complex process. Osteoblasts play an important role during initiation of bone resorption.

Changes OPG expression of osteoblasts under mechanical stimulation can play a role in bone remodeling. In order to test this hypothesis, the following specific aims will be achieved:

1. To test whether levels of OPG can be changed during orthodontic treatment. Alveolar bone samples will be collected from partially impacted third molars after orthodontic uprighting for different period of time in volunteers. In situ hybridization and immunohistochemistry analysis for OPG and RANKL will reveal their roles in this physiological process.
2. To optimize the regulation by changing magnitude and frequency of pressure, and characterize the time table for these changes..

ELIGIBILITY:
Inclusion Criteria:

* patients with two mandibular impaction third molars containing at least one mesially angular impaction with crown exposed to the oral cavity

Exclusion Criteria:

* pregnancy or diseases with abnormal bone metabolism

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
OPG staining | at most 7 days
  at 1, 3, 7 days after orthodontic force application on wisdom teeth, bone covering the tooth will be removed before taking the wisdom tooth out. The tissue section of the bone will be done with immunocytochemistry after de-calicification.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chen Yao, DDS, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Dentistry, National Taiwan University Hospital, Taipei, Taiwan